CLINICAL TRIAL: NCT00434304
Title: Clinical Evaluation of Ropinirole PR/XR Tablets in Monotherapy for Parkinson's Disease - an Open-Label, Uncontrolled Study -
Brief Title: Clinical Evaluation of Ropinirole PR/XR Tablets in Monotherapy for Parkinson's Disease (PD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ROP106064
Record Dates: First submitted 2007-02-09; First posted 2007-02-13 (Estimated); Results first posted 2009-12-23 (Estimated); Last update posted 2018-09-27 (Actual); Status verified 2018-08

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; PD
MeSH Terms: conditions — Parkinson Disease

ARMS (1):
- Ropinirole PR/XR (Experimental)
  Interventions: Drug: Ropinirole prolonged release/extended release(PR/XR)

INTERVENTIONS:
Drug: Ropinirole prolonged release/extended release(PR/XR) — Subjects will take the investigational drug once daily at the same time each day, it is recommended that this is in the morning for optimal benefit. Investigational drug is taken for 52 weeks, starting on the next day of the Week 0 visit. One tablet of ropinirole PR/XR 2 mg tablets will be orally dosed as the initial dose. The dose will be titrated weekly by 2 mg/day, and increased to 8 mg/day in Week 4. From Week 5 up to 16, the dose will be increased at minimum intervals of one week between titration steps until sufficient efficacy is obtained, according to individual clinical response and tolerability (the dose may be titrated up to 16 mg/day). In Week 16 and further, treatment dose at Week 16 will be continuously administered up to Week 52. If insufficient efficacy is judged in a subject during treatment, or unable to maintain the dose due to adverse event, the treatment dose may be changed. The dose is down tapered according to the maintenance dose at Week 52 (or withdrawal).

SUMMARY:
This study was designed to evaluate the pharmacokinetic profile, safety and efficacy in Parkinson's Disease patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed with PD with severity of the Modified Hoehn & Yahr staging at Stage I to III.
* Age: 20 years or older (at the time of giving informed consent)
* Gender: male and female
* Both inpatient and outpatient status
* Informed consent: Patients who are able to give informed written consent in person (i.e. patients who are capable of giving informed written consent on one's own)
* Limited prior exposure to low or moderate doses of L-dopa (up to 3 months in total) or dopamine agonists (up to 6 months in total) provided treatment is discontinued for a minimum of 4 weeks prior to screening.

Exclusion Criteria:

* Patients who present serious physical signs and symptoms other than those of the PD (e.g. cardiac/hepatic/renal disorder and haematopoietic disorder). The seriousness refers to Grade 3 according to "the Classification of the Severity of Adverse Experiences (Pharmaceutical affairs bureau/Safety division (PAB/SD) Notification No. 80, dated 29 June 1992).
* Patients with symptomatic postural hypotension. (e.g. dizziness and syncope).
* Patients who have had serious psychiatric symptoms (e.g. confusion, hallucination, delusion, abnormal behaviour, alcohol or drug dependence) during the past six months (26 weeks) (including symptoms caused by anti-Parkinson drugs).
* Patients who have been treated with the following drugs at Week -4, and whose treatment regimen of the drug has been changed from Week -4 to Week 0.

  * Anticholinergic agents: trihexyphenidyl hydrochloride (e.g. Artane®), piroheptine hydrochloride (Trimol®), mazaticol hydrochloride (Pentona®), metixene hydrochloride (Cholinfall®), biperiden hydrochloride (Akineton®), profenamine (Parkin®)
  * amantadine hydrochloride (e.g. Symmetrel®)
  * droxidopa (Dops®)
  * citicoline (e.g. Nicholin®)
  * selegiline hydrochloride (FP®)
  * zonisamide
  * estrogen: estriol (e.g.Estriel®)
  * CYP1A2 inhibitors: Ciprofloxacin HCl (e.g. Ciproxan®, enoxacin and fluvoxamine)
* Patients with severe dementia such as score 3 or 4 of the UPDRS Part I (Mentation, behaviour, and mood)
* Female patients who are pregnant or lactating, who may be pregnant, or who plan for pregnancy during the study or within 30 days after the last dose of the study drug.
* Patients with current history or complication of carcinoma or malignant tumour.
* Patients who have history of drug allergy to ropinirole hydrochloride (HCl).
* Patients who have received surgical treatment for PD in the past (e.g. pallidectomy, deep brain stimulation).
* Patients who have been treated with any other investigational drug within 12weeks prior to the treatment phase.
* Others whom the investigator (sub investigator) considers ineligible for the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2007-04-09; Primary Completion 2009-03-01 (Actual); Study Completion 2009-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- Japan (10):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Numakunai
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tokyo

RESULTS

PARTICIPANT FLOW:
Groups:
- Ropinirole PR/XR: Treatment Phase: Fixed titration phase (4 weeks): one tablet of ropinirole PR/XR 2 milligrams (mg) as the initial dose. The dose was titrated weekly by 2 mg/day and was increased to 8 mg/day in Week 4; Flexible titration and maintenance dose phases (48 weeks): from Week 5 up to Week 16, the dose was increased at minimum intervals of 1 week between titration steps (up to 16 mg/day). From Week 16 onward, treatment dose was continuously administered up to Week 52. Taper phase: the dose was tapered over 2 to 3 weeks according to the maintenance dose at completion of the Treatment Phase (or withdrawal)
Period: Overall Study
Arm/Group | Ropinirole PR/XR
Started | 62
Completed | 42
Not Completed | 20
Not completed — Adverse Event | 14
Not completed — Lack of Efficacy | 2
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Ropinirole PR/XR
Number analyzed (Participants) | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (8.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 25
Race/Ethnicity, Customized [Number; unit: participants]
  Asian - Japanese Heritage | 62

OUTCOME MEASURES:

1. Primary Outcome: Food Effects on Cmax and Cmin of SKF101468 (Ropinirole) and Its Metabolites
Description: The dose of SKF101468 and its metabolites was normalized to 1 mg. Blood sampling at steady state up to 24 hours post dose after receiving the maintenance dose was conducted. In order to investigate the effect of a meal on pharmacokinetics, blood was sampled twice (after a standard morning meal and at fasted state) from identical participants. Cmax: maximum concentration, Cmin: trough plasma concentration.
Time Frame: Weeks 5-16
Population: Pharmacokinetic (PK) Population: participants who underwent blood sampling for PK research, excluding those who did not fulfill inclusion criteria and those who were considered to affect the evaluation of the PK research due to drug incompliance or other protocol violation.
Measure: Geometric Mean (95% Confidence Interval); unit: picograms/milliliter (pg/mL)
Arm/Group | Ropinirole PR/XR
Number analyzed (Participants) | 10
picograms/milliliter (pg/mL)
  SKF101468 (ropinirole), Cmax, fed | 1563.784 [1252.648 to 1952.202]
  SKF101468 (ropinirole), Cmax, fasted | 1542.182 [1177.843 to 2019.221]
  SKF101468 (ropinirole), Cmin, fed | 728.404 [565.589 to 938.087]
  SKF101468 (ropinirole), Cmin, fasted | 725.103 [546.750 to 961.636]
  SKF104557 (metabolite), Cmax, fed | 1159.120 [1034.646 to 1298.569]
  SKF104557 (metabolite), Cmax, fasted | 1250.554 [1077.255 to 1451.731]
  SKF104557 (metabolite), Cmin, fed | 798.871 [693.490 to 920.266]
  SKF104557 (metabolite), Cmin, fasted | 786.097 [672.811 to 918.458]
  SKF89124 (metabolite), Cmax, fed | 55.282 [46.462 to 65.776]
  SKF89124 (metabolite), Cmax, fasted | 60.742 [48.303 to 76.384]
  SKF89124 (metabolite), Cmin, fed | 34.281 [27.811 to 42.256]
  SKF89124 (metabolite), Cmin, fasted | 34.599 [28.720 to 41.682]

2. Secondary Outcome: Total Score in the Japanese UPDRS Part III
Description: The Unified Parkinson's Disease Rating Scale (UPDRS) assesses the status of Parkinson's Disease (PD) patients objectively. The Japanese UPDRS Part III assesses motor examination on 27 items. Participants receive a score of 0-4 points per each item. The maximum total score is 108 points. A higher score indicates more severe PD symptoms.
Time Frame: Weeks 0-52
Population: Full Analysis Set (FAS): all participants who progressed to the treatment phase, excluding those who did not fulfill major registration criteria, those who had not received at least one dose of the investigational drug, and those whose measured data were not available after treatment initiation. Participants dropped out of the study each week.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Ropinirole PR/XR
Number analyzed (Participants) | 62
points on a scale
  Week 0, n=62 | 22.4 (10.11)
  Week 1, n=62 | 19.3 (9.38)
  Week 2, n=60 | 16.8 (8.89)
  Week 3, n=60 | 14.5 (8.57)
  Week 4, n=58 | 13.0 (8.60)
  Week 6, n=57 | 12.1 (8.47)
  Week 8, n=56 | 11.1 (7.87)
  Week 10, n=57 | 10.2 (7.84)
  Week 12, n=56 | 10.1 (7.18)
  Week 16, n=54 | 10.3 (6.98)
  Final Assessment Point (Up to Week 16), n=62 | 11.1 (7.52)
  Week 20, n=53 | 10.4 (7.20)
  Week 24, n=51 | 10.6 (7.47)
  Week 28, n=48 | 10.6 (7.69)
  Week 32, n=47 | 10.7 (7.68)
  Week 36, n=47 | 10.7 (7.35)
  Week 40, n=45 | 11.0 (8.04)
  Week 44, n=45 | 11.3 (9.30)
  Week 48, n=44 | 10.2 (7.52)
  Week 52, n=44 | 10.7 (7.73)

3. Secondary Outcome: Change From Baseline in the Japanese UPDRS Part III
Description: The UPDRS assesses the status of PD patients objectively. The Japanese UPDRS Part III assesses motor examination on 27 items. Participants receive a score of 0-4 points per each item. The maximum total score is 108 points. A higher score indicates more severe PD symptoms.
Time Frame: Baseline (Week 0) and Weeks 1-52
Population: FAS. Participants dropped out of the study each week.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Ropinirole PR/XR
Number analyzed (Participants) | 62
points on a scale
  Week 1, n=62 | -3.1 (4.21)
  Week 2, n=60 | -5.8 (5.18)
  Week 3, n=60 | -7.7 (6.67)
  Week 4, n=58 | -9.7 (6.77)
  Week 6, n=57 | -10.5 (7.31)
  Week 8, n=56 | -11.5 (7.95)
  Week 10, n=57 | -12.4 (7.57)
  Week 12, n=56 | -12.3 (7.47)
  Week 16, n=54 | -12.2 (8.10)
  Final Assessment Point (Up to Week 16), n=62 | -11.3 (8.21)
  Week 20, n=53 | -12.1 (8.65)
  Week 24, n=51 | -11.6 (8.21)
  Week 28, n=48 | -11.5 (9.04)
  Week 32, n=47 | -11.7 (8.27)
  Week 36, n=47 | -11.7 (8.37)
  Week 40, n=45 | -11.5 (8.26)
  Week 44, n=45 | -11.2 (9.12)
  Week 48, n=44 | -11.9 (8.57)
  Week 52, n=44 | -11.4 (8.55)

4. Secondary Outcome: Percent Change From Baseline in the Japanese UPDRS Part III
Description: The UPDRS assesses the status of PD patients objectively. The Japanese UPDRS Part III assesses motor examination on 27 items. Participants receive a score of 0-4 points per each item. A maximum total score is 108 points.The higher score indicates more severe PD symptoms.
Time Frame: Baseline (Week 0) and Weeks 1-52
Population: FAS. Participants dropped out of the study each week.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ropinirole PR/XR
Number analyzed (Participants) | 62
percent change
  Week 1, n=62 | -14.14 (17.734)
  Week 2, n=60 | -27.14 (23.525)
  Week 3, n=60 | -35.13 (28.125)
  Week 4, n=58 | -45.03 (24.055)
  Week 6, n=57 | -48.35 (26.605)
  Week 8, n=56 | -51.34 (30.203)
  Week 10, n=57 | -56.63 (26.249)
  Week 12, n=56 | -56.24 (23.382)
  Week 16, n=54 | -53.78 (28.309)
  Final Assessment Point (Up to Week 16), n=62 | -49.38 (32.041)
  Week 20, n=53 | -52.61 (32.017)
  Week 24, n=51 | -51.56 (28.676)
  Week 28, n=48 | -50.25 (30.813)
  Week 32, n=47 | -51.67 (26.037)
  Week 36, n=47 | -51.36 (27.300)
  Week 40, n=45 | -50.58 (25.887)
  Week 44, n=45 | -49.51 (32.903)
  Week 48, n=44 | -53.05 (28.456)
  Week 52, n=44 | -51.11 (31.617)

5. Secondary Outcome: Percentage of Responders of the Total Score in the Japanese UPDRS Total Score in Part III
Description: A responder is defined as a participant with a 30% or more reduction at baseline. The UPDRS assesses the status of PD patients objectively. The Japanese UPDRS Part III assesses motor examination on 27 items. Participants receive a score of 0-4 points per each item. The maximum total score is 108 points. A higher score indicates more severe PD symptoms.
Time Frame: Baseline (Week 0) and Weeks 1-52
Population: FAS. Participants dropped out of the study each week.
Measure: Number; unit: percentage of responders
Arm/Group | Ropinirole PR/XR
Number analyzed (Participants) | 62
percentage of responders
  Week 1, n=62 | 12.9
  Week 2, n=60 | 38.3
  Week 3, n=60 | 58.3
  Week 4, n=58 | 70.7
  Week 6, n=57 | 71.9
  Week 8, n=56 | 82.1
  Week 10, n=57 | 84.2
  Week 12, n=56 | 89.3
  Week 16, n=54 | 81.5
  Final Assessment Point (Up to Week 16), n=62 | 75.8
  Week 20, n=53 | 81.1
  Week 24, n=51 | 78.4
  Week 28, n=48 | 79.2
  Week 32, n=47 | 76.6
  Week 36, n=47 | 76.6
  Week 40, n=45 | 77.8
  Week 44, n=45 | 77.8
  Week 48, n=44 | 81.8
  Week 52, n=44 | 81.8

6. Secondary Outcome: Total Score in the Japanese UPDRS Part I
Description: The UPDRS assesses the status of PD patients objectively. The Japanese UPDRS Part I assesses mentation, behavior, and mood on 4 items. Participants receive a score of 0-4 points per each item. The maximum total score is 16 points. A higher score indicates more severe mental symptoms.
Time Frame: Weeks 0-52
Population: FAS. Participants dropped out of the study each week.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Ropinirole PR/XR
Number analyzed (Participants) | 62
points on a scale
  Week 0, n=62 | 1.0 (1.36)
  Week 1, n=62 | 0.7 (1.09)
  Week 2, n=60 | 0.6 (0.96)
  Week 3, n=60 | 0.5 (1.06)
  Week 4, n=58 | 0.4 (1.06)
  Week 6, n=57 | 0.5 (1.04)
  Week 8, n=56 | 0.5 (1.10)
  Week 10, n=57 | 0.6 (1.39)
  Week 12, n=56 | 0.4 (1.07)
  Week 16, n=54 | 0.4 (1.31)
  Final Assessment Point (Up to Week 16), n=62 | 0.4 (1.30)
  Week 20, n=53 | 0.3 (0.88)
  Week 24, n=51 | 0.4 (0.87)
  Week 28, n=48 | 0.3 (0.57)
  Week 32, n=47 | 0.3 (0.61)
  Week 36, n=47 | 0.4 (0.64)
  Week 40, n=45 | 0.3 (0.58)
  Week 44, n=45 | 0.3 (0.67)
  Week 48, n=44 | 0.3 (0.73)
  Week 52, n=44 | 0.3 (0.80)

7. Secondary Outcome: Change From Baseline in the Japanese UPDRS Part I
Description: The UPDRS (Unified Parkinson's Disease Rating Scale) assesses the status of PD patients objectively. The Japanese UPDRS Part I assesses mentation, behavior, and mood on 4 items. Participants receive a score of 0-4 points per each item. The maximum total score is 16 points. A higher score indicates more severe mental symptoms.
Time Frame: Baseline (Week 0) and Weeks 1-52
Population: FAS. Participants dropped out of the study each week.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Ropinirole PR/XR
Number analyzed (Participants) | 62
points on a scale
  Week 1, n=62 | -0.3 (1.00)
  Week 2, n=60 | -0.5 (0.91)
  Week 3, n=60 | -0.5 (1.14)
  Week 4, n=58 | -0.5 (1.13)
  Week 6, n=57 | -0.5 (1.21)
  Week 8, n=56 | -0.5 (1.16)
  Week 10, n=57 | -0.3 (1.21)
  Week 12, n=56 | -0.5 (1.14)
  Week 16, n=54 | -0.6 (1.24)
  Final Assessment Point (Up to Week 16), n=62 | -0.5 (1.21)
  Week 20, n=53 | -0.5 (1.15)
  Week 24, n=51 | -0.5 (1.10)
  Week 28, n=48 | -0.5 (1.11)
  Week 32, n=47 | -0.5 (1.20)
  Week 36, n=47 | -0.4 (1.28)
  Week 40, n=45 | -0.4 (1.16)
  Week 44, n=45 | -0.4 (1.25)
  Week 48, n=44 | -0.4 (1.30)
  Week 52, n=44 | -0.4 (1.30)

8. Secondary Outcome: Percent Change From Baseline in the Japanese UPDRS Part I
Description: as for outcome 7
Time Frame: Baseline (Week 0) and Weeks 1-52
Population: FAS. Participants dropped out of the study each week.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ropinirole PR/XR
Number analyzed (Participants) | 62
percent change
  Week 1, n=30 | -34.17 (48.460)
  Week 2, n=29 | -54.60 (46.269)
  Week 3, n=29 | -63.79 (49.815)
  Week 4, n=28 | -60.71 (49.735)
  Week 6, n=27 | -69.44 (48.205)
  Week 8, n=27 | -54.94 (59.524)
  Week 10, n=27 | -48.46 (66.105)
  Week 12, n=26 | -62.50 (67.956)
  Week 16, n=24 | -77.08 (48.358)
  Final Assessment Point (Up to Week 16), n=30 | -68.89 (52.838)
  Week 20, n=23 | -71.74 (51.354)
  Week 24, n=22 | -65.91 (44.089)
  Week 28, n=20 | -71.67 (50.466)
  Week 32, n=19 | -67.54 (71.465)
  Week 36, n=19 | -55.26 (66.447)
  Week 40, n=17 | -69.61 (55.664)
  Week 44, n=17 | -52.94 (69.531)
  Week 48, n=16 | -59.38 (71.224)
  Week 52, n=16 | -53.13 (71.807)

9. Secondary Outcome: Total Score in the Japanese UPDRS Part II
Description: The UPDRS assesses the status of PD patients objectively. The Japanese UPDRS Part II assesses activities of daily living on 13 items. Participants receive a score of 0-4 points per each item. The maximum total score is 52 points. A higher score indicates more severe PD symptoms.
Time Frame: Weeks 0-52
Population: FAS. Participants dropped out of the study each week.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Ropinirole PR/XR
Number analyzed (Participants) | 62
points on a scale
  Week 0, n=62 | 8.2 (4.55)
  Week 1, n=62 | 7.2 (4.41)
  Week 2, n=60 | 6.3 (4.00)
  Week 3, n=60 | 5.5 (3.82)
  Week 4, n=58 | 4.8 (3.79)
  Week 6, n=57 | 4.5 (3.76)
  Week 8, n=56 | 4.0 (3.64)
  Week 10, n=57 | 4.1 (3.95)
  Week 12, n=56 | 4.2 (3.77)
  Week 16, n=54 | 4.1 (3.50)
  Final Assessment Point (Up to Week 16), n=62 | 4.3 (3.69)
  Week 20, n=53 | 4.1 (3.57)
  Week 24, n=51 | 3.7 (3.38)
  Week 28, n=48 | 4.0 (3.79)
  Week 32, n=47 | 3.9 (3.61)
  Week 36, n=47 | 4.0 (3.73)
  Week 40, n=45 | 4.1 (3.90)
  Week 44, n=45 | 4.2 (4.14)
  Week 48, n=44 | 3.8 (3.88)
  Week 52, n=44 | 4.1 (4.13)

10. Primary Outcome: Food Effects on AUC0-24 of SKF101468 (Ropinirole) and Its Metabolites
Description: The dose of SKF101468 and its metabolites was normalized to 1 mg. Blood sampling at steady state up to 24 hours (hr) post dose after receiving the maintenance dose was conducted. In order to investigate the effect of a meal on pharmacokinetics, blood was sampled twice (after a standard morning meal and at fasted state) from identical participants. AUC0-24: area under the drug concentration 24 hr curve.
Time Frame: Weeks 5-16
Population: PK Population
Measure: Geometric Mean (95% Confidence Interval); unit: hours*pg/mL
Arm/Group | Ropinirole PR/XR
Number analyzed (Participants) | 10
hours*pg/mL
  SKF101468 (ropinirole), fed | 27206.103 [21908.900 to 33784.080]
  SKF101468 (ropinirole), fasted | 27191.804 [20738.729 to 35652.821]
  SKF104557 (metabolite), fed | 23090.150 [20629.318 to 25844.530]
  SKF104557 (metabolite), fasted | 24478.797 [21280.201 to 28158.169]
  SKF89124 (metabolite), fed | 1044.877 [882.879 to 1236.601]
  SKF89124 (metabolite), fasted | 1092.635 [888.375 to 1343.860]

11. Primary Outcome: Food Effects on Tmax of SKF101468 (Ropinirole) and Its Metabolites
Description: The dose of SKF101468 and its metabolites was normalized to 1 mg. Blood sampling at steady state up to 24 hours post dose after receiving the maintenance dose was conducted. In order to investigate the effect of a meal on pharmacokinetics, blood was sampled twice (after a standard morning meal and at fasted state) from identical participants. Tmax: time of maximum concentration. Data are presented as the median difference between fed and fasted states for ropinirole and each metabolite.
Time Frame: Weeks 5-16
Population: PK Population
Measure: Median (90% Confidence Interval); unit: hours
Arm/Group | Ropinirole PR/XR
Number analyzed (Participants) | 10
hours
  SKF101468 (ropinirole) | 2.000 [-0.100 to 5.000]
  SKF104557 (metabolite) | 3.983 [2.000 to 6.000]
  SKF89124 (metabolite) | 1.000 [-0.100 to 5.000]

12. Primary Outcome: Plasma Trough Concentrations of SKF101468 (Ropinirole) and Its Metabolites
Description: Blood sampling in the fixed titration phase will be performed at 24 hour post dose of the last dose of 2, 4, and 8 mg (immediately before the morning dose). Blood sampling in the maintenance dose phase will be performed at 24 hour post dose of 10 mg or more for one week or longer (immediately before the morning dose), as sampling needs to be conducted at steady state.
Time Frame: Weeks 1-16
Population: PK Population. Blood sampling was performed in all participants in the Fixed titration phase and Maintenance dose phase to measure trough concentration. The maintenance dose differs for individual participants.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Ropinirole PR/XR
Number analyzed (Participants) | 61
pg/mL
  SKF101468 (ropinirole), 2 mg, n=61 | 1804.87 (1757.062)
  SKF101468 (ropinirole), 4 mg, n=58 | 3529.59 (1746.855)
  SKF101468 (ropinirole), 6 mg, n=1 | 3820.20 (0.000)
  SKF101468 (ropinirole), 8 mg, n=61 | 7598.90 (5512.105)
  SKF101468 (ropinirole), 10 mg, n=17 | 9772.23 (3237.589)
  SKF101468 (ropinirole), 12 mg, n=12 | 11971.49 (7211.987)
  SKF101468 (ropinirole), 14 mg, n=9 | 12575.41 (5586.121)
  SKF101468 (ropinirole), 16 mg, n=12 | 15467.01 (8292.375)
  SKF104557 (metabolite), 2 mg, n=61 | 1564.52 (777.387)
  SKF104557 (metabolite), 4 mg, n=58 | 3224.53 (1184.861)
  SKF104557 (metabolite), 6 mg, n=1 | 4172.10 (0.000)
  SKF104557 (metabolite), 8 mg, n=61 | 6353.30 (2173.457)
  SKF104557 (metabolite), 10 mg, n=17 | 7944.70 (1887.958)
  SKF104557 (metabolite), 12 mg, n=12 | 11814.28 (3917.886)
  SKF104557 (metabolite), 14 mg, n=9 | 11579.79 (4279.464)
  SKF104557 (metabolite), 16 mg, n=12 | 12753.83 (2527.639)
  SKF89124 (metabolite), 2 mg, n=61 | 66.14 (39.824)
  SKF89124 (metabolite), 4 mg, n=58 | 139.84 (56.099)
  SKF89124 (metabolite), 6 mg, n=1 | 157.40 (0.000)
  SKF89124 (metabolite), 8 mg, n=61 | 281.36 (120.381)
  SKF89124 (metabolite), 10 mg, n=17 | 318.82 (83.774)
  SKF89124 (metabolite), 12 mg, n=12 | 479.36 (189.388)
  SKF89124 (metabolite), 14 mg, n=9 | 564.57 (286.257)
  SKF89124 (metabolite), 16 mg, n=12 | 628.76 (271.495)

13. Secondary Outcome: Change From Baseline in the Japanese UPDRS Part II
Description: as for outcome 9
Time Frame: Baseline (Week 0) and Weeks 1-52
Population: FAS. Participants dropped out of the study each week.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Ropinirole PR/XR
Number analyzed (Participants) | 62
points on a scale
  Week 1, n=62 | -1.0 (1.60)
  Week 2, n=60 | -1.9 (2.14)
  Week 3, n=60 | -2.6 (2.44)
  Week 4, n=58 | -3.4 (2.84)
  Week 6, n=57 | -3.7 (2.74)
  Week 8, n=56 | -4.2 (3.09)
  Week 10, n=57 | -4.1 (3.16)
  Week 12, n=56 | -4.0 (3.20)
  Week 16, n=54 | -4.1 (3.28)
  Final Assessment Point (Up to Week 16), n=62 | -3.9 (3.22)
  Week 20, n=53 | -4.1 (3.50)
  Week 24, n=51 | -4.4 (3.48)
  Week 28, n=48 | -4.0 (3.75)
  Week 32, n=47 | -4.2 (3.66)
  Week 36, n=47 | -4.1 (3.80)
  Week 40, n=45 | -3.9 (3.98)
  Week 44, n=45 | -3.8 (3.84)
  Week 48, n=44 | -4.0 (3.96)
  Week 52, n=44 | -3.7 (4.42)

14. Secondary Outcome: Percent Change From Baseline in the Japanese UPDRS Part II
Description: as for outcome 9
Time Frame: Baseline (Week 0) and Weeks 1-52
Population: FAS. Participants dropped out of the study each week.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ropinirole PR/XR
Number analyzed (Participants) | 62
percent change
  Week 1, n=60 | -11.01 (20.504)
  Week 2, n=58 | -23.04 (26.252)
  Week 3, n=58 | -33.09 (26.531)
  Week 4, n=56 | -44.30 (28.348)
  Week 6, n=55 | -48.89 (28.058)
  Week 8, n=54 | -53.88 (29.274)
  Week 10, n=55 | -52.52 (35.133)
  Week 12, n=54 | -51.51 (31.572)
  Week 16, n=52 | -50.78 (35.826)
  Final Assessment Point (Up to Week 16), n=60 | -49.03 (35.664)
  Week 20, n=51 | -50.10 (35.694)
  Week 24, n=49 | -54.29 (31.096)
  Week 28, n=46 | -51.15 (35.620)
  Week 32, n=45 | -50.91 (37.745)
  Week 36, n=45 | -51.05 (35.493)
  Week 40, n=43 | -48.31 (41.477)
  Week 44, n=43 | -47.48 (40.194)
  Week 48, n=42 | -49.28 (38.285)
  Week 52, n=42 | -41.48 (48.287)

15. Secondary Outcome: Total Score in the Japanese UPDRS Part IV
Description: The UPDRS assesses the status of PD patients objectively. The Japanese UPDRS Part IV assesses complications of therapy on 11 items. Participants receive a score of 0-4 or 0-1 points per each item depending on the item. The maximum total score is 23 points. A higher score indicates more severe symptoms of complications.
Time Frame: Baseline (Week 0) and Weeks 0-52
Population: FAS. Participants dropped out of the study each week.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Ropinirole PR/XR
Number analyzed (Participants) | 62
points on a scale
  Week 0, n=62 | 0.4 (0.58)
  Week 1, n=62 | 0.6 (0.71)
  Week 2, n=60 | 0.8 (0.82)
  Week 3, n=60 | 0.7 (0.78)
  Week 4, n=58 | 0.7 (0.82)
  Week 6, n=57 | 0.7 (0.78)
  Week 8, n=56 | 0.5 (0.63)
  Week 10, n=57 | 0.5 (0.68)
  Week 12, n=56 | 0.5 (0.66)
  Week 16, n=54 | 0.6 (0.63)
  Final Assessment Point (Up to Week 16), n=62 | 0.6 (0.66)
  Week 20, n=53 | 0.6 (0.71)
  Week 24, n=51 | 0.5 (0.64)
  Week 28, n=48 | 0.6 (0.70)
  Week 32, n=47 | 0.5 (0.62)
  Week 36, n=47 | 0.6 (0.62)
  Week 40, n=45 | 0.4 (0.58)
  Week 44, n=45 | 0.5 (0.59)
  Week 48, n=44 | 0.5 (0.59)
  Week 52, n=44 | 0.5 (0.63)

16. Secondary Outcome: Change From Baseline in the Japanese UPDRS Part IV
Description: as for outcome 15
Time Frame: Baseline (Week 0) and Weeks 1-52
Population: FAS. Participants dropped out of the study each week.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Ropinirole PR/XR
Number analyzed (Participants) | 62
points on a scale
  Week 1, n=62 | 0.2 (0.64)
  Week 2, n=60 | 0.4 (0.74)
  Week 3, n=60 | 0.3 (0.74)
  Week 4, n=58 | 0.3 (0.78)
  Week 6, n=57 | 0.3 (0.83)
  Week 8, n=56 | 0.2 (0.74)
  Week 10, n=57 | 0.2 (0.70)
  Week 12, n=56 | 0.2 (0.72)
  Week 16, n=54 | 0.2 (0.63)
  Final Assessment Point (Up to Week 16), n=62 | 0.2 (0.66)
  Week 20, n=53 | 0.3 (0.67)
  Week 24, n=51 | 0.2 (0.68)
  Week 28, n=48 | 0.3 (0.75)
  Week 32, n=47 | 0.2 (0.70)
  Week 36, n=47 | 0.3 (0.71)
  Week 40, n=45 | 0.1 (0.66)
  Week 44, n=45 | 0.2 (0.63)
  Week 48, n=44 | 0.3 (0.72)
  Week 52, n=44 | 0.2 (0.74)

17. Secondary Outcome: Percent Change From Baseline in the Japanese UPDRS Part IV
Description: as for outcome 15
Time Frame: Baseline (Week 0) and Weeks 1-52
Population: FAS. Participants dropped out of the study each week.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ropinirole PR/XR
Number analyzed (Participants) | 62
percent change
  Week 1, n=21 | -2.38 (64.180)
  Week 2, n=20 | 17.50 (71.221)
  Week 3, n=19 | 10.53 (79.196)
  Week 4, n=19 | 7.89 (75.024)
  Week 6, n=18 | -5.56 (72.536)
  Week 8, n=17 | -35.29 (60.634)
  Week 10, n=18 | -16.67 (70.711)
  Week 12, n=17 | -14.71 (70.189)
  Week 16, n=16 | -15.63 (50.724)
  Final Assessment Point (Up to Week 16), n=21 | -16.67 (48.305)
  Week 20, n=15 | -6.67 (79.881)
  Week 24, n=14 | -25.00 (58.012)
  Week 28, n=13 | -23.08 (59.914)
  Week 32, n=13 | -34.62 (62.532)
  Week 36, n=13 | -26.92 (72.501)
  Week 40, n=12 | -41.67 (79.296)
  Week 44, n=12 | -25.00 (75.378)
  Week 48, n=12 | -41.67 (66.856)
  Week 52, n=12 | -41.67 (51.493)

18. Secondary Outcome: Summary of the Modified Hoehn & Yahr Criteria Stages
Description: Hoehn & Yahr criteria were measured on an 8-point scale. 0: No signs of disease, 1: Unilateral disease, 1.5: Unilateral plus axial involvement, 2: Bilateral disease, 2.5: Mild bilateral disease, 3: Mild to moderate bilateral disease. No subjects evaluated had a score of 4 (severe disability) or 5 (wheelchair bound or bedridden unless aided).
Time Frame: Screening-Week 52
Population: FAS. Participants dropped out of the study each week.
Measure: Number; unit: points on a scale
Arm/Group | Ropinirole PR/XR
Number analyzed (Participants) | 62
points on a scale
  Screening, Stage 0 | 0
  Screening, Stage 1 | 7
  Screening, Stage 1.5 | 7
  Screening, Stage 2 | 18
  Screening, Stage 2.5 | 12
  Screening, Stage 3 | 18
  Week 0, Stage 0 | 0
  Week 0, Stage 1 | 6
  Week 0, Stage 1.5 | 5
  Week 0, Stage 2 | 23
  Week 0, Stage 2.5 | 12
  Week 0, Stage 3 | 16
  Week 1, Stage 0 | 0
  Week 1, Stage 1 | 8
  Week 1, Stage 1.5 | 4
  Week 1, Stage 2 | 24
  Week 1, Stage 2.5 | 12
  Week 1, Stage 3 | 14
  Week 2, Stage 0 | 1
  Week 2, Stage 1 | 8
  Week 2, Stage 1.5 | 5
  Week 2, Stage 2 | 22
  Week 2, Stage 2.5 | 12
  Week 2, Stage 3 | 12
  Week 3, Stage 0 | 0
  Week 3, Stage 1 | 12
  Week 3, Stage 1.5 | 3
  Week 3, Stage 2 | 26
  Week 3, Stage 2.5 | 8
  Week 3, Stage 3 | 11
  Week 4, Stage 0 | 0
  Week 4, Stage 1 | 12
  Week 4, Stage 1.5 | 5
  Week 4, Stage 2 | 26
  Week 4, Stage 2.5 | 7
  Week 4, Stage 3 | 8
  Week 6, Stage 0 | 1
  Week 6, Stage 1 | 17
  Week 6, Stage 1.5 | 4
  Week 6, Stage 2 | 23
  Week 6, Stage 2.5 | 3
  Week 6, Stage 3 | 9
  Week 8, Stage 0 | 1
  Week 8, Stage 1 | 18
  Week 8, Stage 1.5 | 5
  Week 8, Stage 2 | 21
  Week 8, Stage 2.5 | 7
  Week 8, Stage 3 | 4
  Week 10, Stage 0 | 3
  Week 10, Stage 1 | 19
  Week 10, Stage 1.5 | 7
  Week 10, Stage 2 | 21
  Week 10, Stage 2.5 | 2
  Week 10, Stage 3 | 5
  Week 12, Stage 0 | 3
  Week 12, Stage 1 | 18
  Week 12, Stage 1.5 | 8
  Week 12, Stage 2 | 17
  Week 12, Stage 2.5 | 5
  Week 12, Stage 3 | 5
  Week 16, Stage 0 | 3
  Week 16, Stage 1 | 16
  Week 16, Stage 1.5 | 6
  Week 16, Stage 2 | 20
  Week 16, Stage 2.5 | 4
  Week 16, Stage 3 | 5
  Final Assessment Point (Up to Week 16), Stage 0 | 3
  Final Assessment Point (Up to Week 16), Stage 1 | 18
  Final Assessment Point (Up to Week 16), Stage 1.5 | 6
  Final Assessment Point (Up to Week 16), Stage 2 | 23
  Final Assessment Point (Up to Week 16), Stage 2.5 | 5
  Final Assessment Point (Up to Week 16), Stage 3 | 7
  Week 20, Stage 0 | 4
  Week 20, Stage 1 | 16
  Week 20, Stage 1.5 | 3
  Week 20, Stage 2 | 20
  Week 20, Stage 2.5 | 3
  Week 20, Stage 3 | 7
  Week 24, Stage 0 | 3
  Week 24, Stage 1 | 14
  Week 24, Stage 1.5 | 3
  Week 24, Stage 2 | 22
  Week 24, Stage 2.5 | 4
  Week 24, Stage 3 | 5
  Week 28, Stage 0 | 2
  Week 28, Stage 1 | 14
  Week 28, Stage 1.5 | 4
  Week 28, Stage 2 | 17
  Week 28, Stage 2.5 | 5
  Week 28, Stage 3 | 6
  Week 32, Stage 0 | 2
  Week 32, Stage 1 | 14
  Week 32, Stage 1.5 | 2
  Week 32, Stage 2 | 19
  Week 32, Stage 2.5 | 5
  Week 32, Stage 3 | 5
  Week 36, Stage 0 | 2
  Week 36, Stage 1 | 13
  Week 36, Stage 1.5 | 2
  Week 36, Stage 2 | 19
  Week 36, Stage 2.5 | 6
  Week 36, Stage 3 | 5
  Week 40, Stage 0 | 2
  Week 40, Stage 1 | 12
  Week 40, Stage 1.5 | 2
  Week 40, Stage 2 | 18
  Week 40, Stage 2.5 | 7
  Week 40, Stage 3 | 4
  Week 44, Stage 0 | 2
  Week 44, Stage 1 | 16
  Week 44, Stage 1.5 | 2
  Week 44, Stage 2 | 14
  Week 44, Stage 2.5 | 5
  Week 44, Stage 3 | 6
  Week 48, Stage 0 | 1
  Week 48, Stage 1 | 16
  Week 48, Stage 1.5 | 1
  Week 48, Stage 2 | 16
  Week 48, Stage 2.5 | 4
  Week 48, Stage 3 | 6
  Week 52, Stage 0 | 1
  Week 52, Stage 1 | 15
  Week 52, Stage 1.5 | 2
  Week 52, Stage 2 | 16
  Week 52, Stage 2.5 | 5
  Week 52, Stage 3 | 5

19. Secondary Outcome: Number of Participants Scored as Responders on the Clinician's Global Impression (CGI) Scale
Description: CGI is measured on a 7-point scale. 1: Very much improved, 2: Much Improved, 3: Minimally improved, 4: No change, 5: Minimally worse, 6: Much worse, 7: Very much worse. Responders are defined as those participants scored as "very much improved" or "much improved."
Time Frame: Weeks 1-52
Population: FAS. Participants dropped out of the study each week.
Measure: Number; unit: participants
Arm/Group | Ropinirole PR/XR
Number analyzed (Participants) | 62
participants
  Week 1, n=62 | 8
  Week 2, n=60 | 16
  Week 3, n=60 | 25
  Week 4, n=58 | 39
  Week 6, n=57 | 40
  Week 8, n=56 | 45
  Week 10, n=57 | 47
  Week 12, n=56 | 48
  Week 16, n=54 | 41
  Final Assessment Point (Up to Week 16), n=62 | 44
  Week 20, n=53 | 43
  Week 24, n=51 | 40
  Week 28, n=48 | 38
  Week 32, n=47 | 35
  Week 36, n=47 | 35
  Week 40, n=45 | 33
  Week 44, n=45 | 35
  Week 48, n=44 | 37
  Week 52, n=44 | 35

20. Secondary Outcome: Percentage of Participants Who Remained in the Study on the Indicated Days
Description: The percentage of participants remaining in the study was examined using the Kaplan-Meier method, in which a premature discontinuation will be considered as an event.
Time Frame: Days 0-364
Population: FAS. Participants dropped out of the study each week.
Measure: Number; unit: percentage of participants
Arm/Group | Ropinirole PR/XR
Number analyzed (Participants) | 62
percentage of participants
  Day 0 | 100
  Day 10 | 98
  Day 14 | 97
  Day 21 | 94
  Day 28 | 92
  Day 70 | 90
  Day 84 | 89
  Day 96 | 87
  Day 112 | 85
  Day 140 | 84
  Day 168 | 82
  Day 175 | 79
  Day 183 | 77
  Day 196 | 76
  Day 239 | 74
  Day 252 | 73
  Day 315 | 71
  Day 359 | 69
  Day 364 | 67

21. Secondary Outcome: Change From Baseline in Albumin, Total Protein, and Hemoglobin at Weeks 16 and 52
Description: Change from baseline was calculated as the Week 16 and 52 values minus the baseline values.
Time Frame: Baseline (Screening) and Weeks 16 and 52
Population: Safety Population: all participants who received at least one dose of study medication. Week 16 (Last observation carried forward [LOCF]) = 62 participants; Week 52 (Observed case [OC]) = 44 participants
Measure: Mean (Standard Deviation); unit: grams per Liter (G/L)
Arm/Group | Ropinirole PR/XR
Number analyzed (Participants) | 62
grams per Liter (G/L)
  Albumin, Week 16 | -0.66 (1.983)
  Albumin, Week 52 | -1.68 (2.428)
  Total Protein, Week 16 | -1.71 (3.761)
  Total Protein, Week 52 | -2.32 (3.665)
  Hemoglobin, Week 16 | -4.44 (9.557)
  Hemoglobin, Week 52 | -4.00 (11.477)

22. Secondary Outcome: Change From Baseline in Alkaline Phosphatase, Alanine Amino Transferase, Aspartate Amino Transferase, Creatine Kinase, Gamma Glutamyl Transferase, and Lactate Dehydrogenase at Weeks 16 and 52
Description: Change from baseline was calculated as the Week 16 and 52 values minus the baseline values.
Time Frame: Baseline (Screening) and Weeks 16 and 52
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: international units per Liter (IU/L)
Arm/Group | Ropinirole PR/XR
Number analyzed (Participants) | 62
international units per Liter (IU/L)
  Alkaline Phosphatase, Week 16 | 16.5 (47.25)
  Alkaline Phosphatase, Week 52 | 2.5 (37.78)
  Alanine Amino Transferase, Week 16 | 1.1 (9.34)
  Alanine Amino Transferase, Week 52 | 2.3 (13.34)
  Aspartate Amino Transferase, Week 16 | 0.3 (6.71)
  Aspartate Amino Transferase, Week 52 | 2.0 (9.14)
  Creatine Kinase, Week 16 | 5.7 (117.47)
  Creatine Kinase, Week 52 | 44.0 (142.26)
  Gamma Glutamyl transferase, Week 16 | -0.2 (21.60)
  Gamma Glutamyl transferase, Week 52 | -3.6 (28.47)
  Lactate Dehydrogenase, Week 16 | -2.9 (28.59)
  Lactate Dehydrogenase, Week 52 | 8.7 (34.25)

23. Secondary Outcome: Change From Baseline in Total Bilirubin, Blood Urea Nitrogen, and Creatinine at Weeks 16 and 52
Description: Change from baseline was calculated as the Week 16 and 52 values minus the baseline values.
Time Frame: Baseline (Screening) and Weeks 16 and 52
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: micromoles per Liter (UMOL/L)
Arm/Group | Ropinirole PR/XR
Number analyzed (Participants) | 62
micromoles per Liter (UMOL/L)
  Total Bilirubin, Week 16 | 0.19 (3.806)
  Total Bilirubin, Week 52 | 0.12 (2.429)
  Creatinine, Week 16 | 2.281 (6.780)
  Creatinine, Week 52 | 1.266 (7.763)

24. Secondary Outcome: Change From Baseline in Blood Urea Nitrogen, Cholesterol, Chloride, Potassium, and Sodium at Weeks 16 and 52
Description: Change from baseline was calculated as the Week 16 and 52 values minus the baseline values.
Time Frame: Baseline (Screening) and Weeks 16 and 52
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: millimoles per Liter (MMOL/L)
Arm/Group | Ropinirole PR/XR
Number analyzed (Participants) | 62
millimoles per Liter (MMOL/L)
  Blood Urea Nitrogen, Week 16 | 0.02 (1.448)
  Blood Urea Nitrogen, Week 52 | 0.19 (1.512)
  Cholesterol, Week 16 | -0.3 (0.65)
  Cholesterol, Week 52 | -0.3 (0.59)
  Chloride, Week 16 | -0.1 (2.62)
  Chloride, Week 52 | 0.4 (2.13)
  Potassium, Week 16 | -0.01 (0.334)
  Potassium, Week 52 | -0.03 (0.378)
  Sodium, Week 16 | -0.1 (2.46)
  Sodium, Week 52 | -0.1 (1.92)

25. Secondary Outcome: Change From Baseline in Prolactin at Weeks 16 and 52
Description: Change from baseline was calculated as the Week 16 and 52 values minus the baseline values.
Time Frame: Baseline (Screening) and Weeks 16 and 52
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: micrograms per Liter (MCG/L)
Arm/Group | Ropinirole PR/XR
Number analyzed (Participants) | 62
micrograms per Liter (MCG/L)
  Week 16 | -7.22 (7.132)
  Week 52 | -8.18 (2.495)

26. Secondary Outcome: Change From Baseline in Hematocrit at Weeks 16 and 52
Description: Change from baseline was calculated as the Week 16 and 52 values minus the baseline values.
Time Frame: Baseline (Screening) and Weeks 16 and 52
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: proportion of 1 (SI)
Arm/Group | Ropinirole PR/XR
Number analyzed (Participants) | 62
proportion of 1 (SI)
  Week 16 | -0.01 (0.028)
  Week 52 | -0.01 (0.028)

27. Secondary Outcome: Change From Baseline in Platelet Count and White Blood Cell Count at Weeks 16 and 52
Description: Change from baseline was calculated as the Week 16 and 52 values minus the baseline values.
Time Frame: Baseline (Screening) and Weeks 16 and 52
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: giga per Liter (GI/L)
Arm/Group | Ropinirole PR/XR
Number analyzed (Participants) | 62
giga per Liter (GI/L)
  Platelet count, Week 16 | -6.81 (31.618)
  Platelet count, Week 52 | -8.07 (44.229)
  White Blood Cell Count, Week 16 | -0.6 (1.30)
  White Blood Cell Count, Week 52 | -0.5 (1.10)

28. Secondary Outcome: Change From Baseline in Red Blood Cell Count at Weeks 16 and 52
Description: Change from baseline was calculated as the Week 16 and 52 values minus the baseline values.
Time Frame: Baseline (Screening) and Weeks 16 and 52
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: tera per Liter (TI/L)
Arm/Group | Ropinirole PR/XR
Number analyzed (Participants) | 62
tera per Liter (TI/L)
  Week 16 | -0.1 (0.26)
  Week 52 | -0.2 (0.27)

29. Secondary Outcome: Urinalysis Data
Description: The number of participants with the indicated dipstick test values were measured. Dipstick test values: Neg Value, Trace, +1, +2, +3, +4. No participants had a score of +5.
Time Frame: Screening, Week 16, and Week 52
Population: Safety Population: Screening Week 16 (LOCF) = 62 participants; Week 52 (OC) = 44 participants
Measure: Number; unit: participants
Arm/Group | Ropinirole PR/XR
Number analyzed (Participants) | 62
participants
  Urine Occult Blood - Screening: Neg Value | 52
  Urine Occult Blood - Screening: Trace | 7
  Urine Occult Blood - Screening: +1 | 1
  Urine Occult Blood - Screening: +2 | 1
  Urine Occult Blood - Screening: +3 | 1
  Urine Occult Blood - Screening: +4 | 0
  Urine Occult Blood - Week 16: Neg Value | 53
  Urine Occult Blood - Week 16: Trace | 4
  Urine Occult Blood - Week 16: +1 | 5
  Urine Occult Blood - Week 16: +2 | 0
  Urine Occult Blood - Week 16: +3 | 0
  Urine Occult Blood - Week 16: +4 | 0
  Urine Occult Blood - Week 52: Neg Value | 41
  Urine Occult Blood - Week 52: Trace | 1
  Urine Occult Blood - Week 52: +1 | 2
  Urine Occult Blood - Week 52: +2 | 0
  Urine Occult Blood - Week 52: +3 | 0
  Urine Occult Blood - Week 52: +4 | 0
  Urine Glucose - Screening: Neg Value | 57
  Urine Glucose - Screening: Trace | 0
  Urine Glucose - Screening: +1 | 1
  Urine Glucose - Screening: +2 | 2
  Urine Glucose - Screening: +3 | 1
  Urine Glucose - Screening: +4 | 1
  Urine Glucose - Week 16: Neg Value | 59
  Urine Glucose - Week 16: Trace | 0
  Urine Glucose - Week 16: +1 | 2
  Urine Glucose - Week 16: +2 | 0
  Urine Glucose - Week 16: +3 | 0
  Urine Glucose - Week 16: +4 | 1
  Urine Glucose - Week 52: Neg Value | 41
  Urine Glucose - Week 52: Trace | 2
  Urine Glucose - Week 52: +1 | 0
  Urine Glucose - Week 52: +2 | 0
  Urine Glucose - Week 52: +3 | 0
  Urine Glucose - Week 52: +4 | 1
  Urine Protein - Screening: Neg Value | 60
  Urine Protein - Screening: Trace | 0
  Urine Protein - Screening: +1 | 2
  Urine Protein - Screening: +2 | 0
  Urine Protein - Screening: +3 | 0
  Urine Protein - Screening: +4 | 0
  Urine Protein - Week 16: Neg Value | 55
  Urine Protein - Week 16: Trace | 3
  Urine Protein - Week 16: +1 | 3
  Urine Protein - Week 16: +2 | 1
  Urine Protein - Week 16: +3 | 0
  Urine Protein - Week 16: +4 | 0
  Urine Protein - Week 52: Neg Value | 43
  Urine Protein - Week 52: Trace | 0
  Urine Protein - Week 52: +1 | 1
  Urine Protein - Week 52: +2 | 0
  Urine Protein - Week 52: +3 | 0
  Urine Protein - Week 52: +4 | 0
  Urine Urobilinogen - Screening: Neg Value | 0
  Urine Urobilinogen - Screening: Trace | 62
  Urine Urobilinogen - Screening: +1 | 0
  Urine Urobilinogen - Screening: +2 | 0
  Urine Urobilinogen - Screening: +3 | 0
  Urine Urobilinogen - Screening: +4 | 0
  Urine Urobilinogen - Week 16: Neg Value | 0
  Urine Urobilinogen - Week 16: Trace | 61
  Urine Urobilinogen - Week 16: +1 | 1
  Urine Urobilinogen - Week 16: +2 | 0
  Urine Urobilinogen - Week 16: +3 | 0
  Urine Urobilinogen - Week 16: +4 | 0
  Urine Urobilinogen - Week 52: Neg Value | 0
  Urine Urobilinogen - Week 52: Trace | 43
  Urine Urobilinogen - Week 52: +1 | 1
  Urine Urobilinogen - Week 52: +2 | 0
  Urine Urobilinogen - Week 52: +3 | 0
  Urine Urobilinogen - Week 52: +4 | 0

30. Secondary Outcome: Number of Participants With the Indicated Shift From Baseline in 12-Lead Electrocardiogram (ECG) Findings at Weeks 16 and 52
Description: Baseline Finding/Time Period Finding. Abbreviations: N = normal; A = abnormal; CS = clinically significant; NCS = not clinically significant. Options include N/N, N/ANCS, N/ACS, ANCS/N, ANCS/ANCS, ANCS/ACS, ACS/N, ACS/ANCS, and ACS/ACS.
Time Frame: Baseline (Screening) and Weeks 16 and 52
Population: Safety Population: Week 16 (LOCF) = 62 participants; Week 52 (OC) = 44 participants
Measure: Number; unit: participants
Arm/Group | Ropinirole PR/XR
Number analyzed (Participants) | 62
participants
  Baseline: N; Week 16: N | 32
  Baseline: N; Week 16: ANCS | 10
  Baseline: N; Week 16: ACS | 0
  Baseline: ANCS; Week 16: N | 5
  Baseline: ANCS; Week 16: ANCS | 13
  Baseline: ANCS; Week 16: ACS | 0
  Baseline: ACS; Week 16: N | 0
  Baseline: ACS; Week 16: ANCS | 0
  Baseline: ACS; Week 16: ACS | 2
  Baseline: N; Week 52: N | 26
  Baseline: N; Week 52: ANCS | 3
  Baseline: N; Week 52: ACS | 0
  Baseline: ANCS; Week 52: N | 5
  Baseline: ANCS; Week 52: ANCS | 9
  Baseline: ANCS; Week 52: ACS | 0
  Baseline: ACS; Week 52: N | 0
  Baseline: ACS; Week 52: ANCS | 0
  Baseline: ACS; Week 52: ACS | 1

31. Secondary Outcome: Change From Baseline in Supine and Standing Systolic and Diastolic Blood Pressure at Weeks 16 and 52
Description: Change from baseline was calculated as Week 16 and Week 52 values minus baseline values.
Time Frame: Baseline (Screening) and Weeks 16 and 52
Population: Safety Population: Week 16 (LOCF) = 62 participants; Week 52 (OC) = 44 participants
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Ropinirole PR/XR
Number analyzed (Participants) | 62
millimeters of mercury (mmHg)
  Supine Systolic BP - Week 16 | -0.0 (20.54)
  Supine Systolic BP - Week 52 | -1.2 (22.84)
  Supine Diastolic BP - Week 16 | 0.6 (11.57)
  Supine Diastolic BP - Week 52 | -1.2 (12.06)
  Standing Systolic BP - Week 16 | -0.7 (19.77)
  Standing Systolic BP - Week 52 | 0.0 (19.08)
  Standing Diastolic BP - Week 16 | -0.7 (12.93)
  Standing Diastolic BP - Week 52 | 2.1 (12.17)

32. Secondary Outcome: Change From Baseline in Supine and Standing Pulse Rate at Weeks 16 and 52
Description: Change from baseline was calculated as Week 16 and Week 52 values minus baseline values.
Time Frame: Baseline (Screening) and Weeks 16 and 52
Population: Safety Population: Week 16 (LOCF) = 62 participants; Week 52 (OC) = 44 participants
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Ropinirole PR/XR
Number analyzed (Participants) | 62
beats per minute (bpm)
  Supine Heart Rate - Week 16 | 0.2 (9.13)
  Supine Heart Rate - Week 52 | -2.3 (11.22)
  Standing Heart Rate - Week 16 | 0.2 (10.32)
  Standing Heart Rate - Week 52 | 0.0 (9.43)

ADVERSE EVENTS:
Groups:
- Ropinirole PR/XR (Treatment Phase): Fixed titration phase (4 weeks): one tablet of ropinirole PR/XR 2 mg as the initial dose. The dose was titrated weekly by 2 mg/day and was increased to 8 mg/day in Week 4; Flexible titration and maintenance dose phases (48 weeks): from Week 5 up to Week 16, the dose was increased at minimum intervals of 1 week between titration steps (up to 16 mg/day). From Week 16 onward, treatment dose was continuously administered up to Week 52.
- Ropinirole PR/XR (Taper Phase): The dose was tapered over 2 to 3 weeks according to the maintenance dose at completion of the Treatment Phase (or withdrawal)
Arm/Group | Ropinirole PR/XR (Treatment Phase) | Ropinirole PR/XR (Taper Phase)
Serious Adverse Events (participants affected / at risk) | 5/62 | 1/62
Other Adverse Events (participants affected / at risk) | 51/62 | 0/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ropinirole PR/XR (Treatment Phase) (N=62) | Ropinirole PR/XR (Taper Phase) (N=62)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Glomerulonephritis rapidly progressive (Renal and urinary disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ropinirole PR/XR (Treatment Phase) (N=62) | Ropinirole PR/XR (Taper Phase) (N=62)
Nausea (Gastrointestinal disorders) | 18 | 0
Constipation (Gastrointestinal disorders) | 16 | 0
Vomiting (Gastrointestinal disorders) | 5 | 0
Stomach discomfort (Gastrointestinal disorders) | 4 | 0
Somnolence (Nervous system disorders) | 25 | 0
Dizziness (Nervous system disorders) | 5 | 0
Headache (Nervous system disorders) | 5 | 0
Hallucination (Psychiatric disorders) | 13 | 0
Nasopharyngitis (Infections and infestations) | 12 | 0
Bronchitis (Infections and infestations) | 4 | 0
Edema peripheral (General disorders) | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.